CLINICAL TRIAL: NCT01719458
Title: Norepinephrine Transporter Imaging in Addiction Disorders
Status: Withdrawn | Type: Observational
Sponsor: Yale University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Marc Potenza, Professor of Psychiatry, Child Study, and Neurobiology, Yale University
Other Study IDs: 0705002688; RL1AA017540 (NIH)
Record Dates: First submitted 2012-10-29; First posted 2012-11-01 (Estimated); Last update posted 2023-03-02 (Actual); Status verified 2023-03

CONDITIONS: Obesity; Alcohol Dependence
MeSH Terms: conditions — Obesity; Alcoholism | interventions — O-methyl reboxetine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Alcohol: Subjects diagnosed with alcohol dependence
  Interventions: Drug: (S,S)-[11C]MRB
- Obese: Subjects diagnosed with obesity
  Interventions: Drug: (S,S)-[11C]MRB
- Healthy: Subjects deemed to be medically healthy
  Interventions: Drug: (S,S)-[11C]MRB

INTERVENTIONS:
Drug: (S,S)-[11C]MRB — PET radioligand

SUMMARY:
In this study we propose to study 24 unmedicated abstinent alcohol dependent patients, 24 obese individuals and 24 individually matched healthy control subjects and determine Norepinephrine Transporter (NET) expression in vivo using (S,S)-[11C]MRB and PET.

DETAILED DESCRIPTION:
In this study we propose to study 24 unmedicated abstinent alcohol dependent patients, 24 obese individuals and 24 individually matched healthy control subjects and determine NET expression in vivo using (S,S)-[11C]MRB and PET. This will provide novel insight into alterations in pre- and post-synaptic homeostasis in alcoholism and obese people with the goal to explain regulatory processes and their alterations in these disorders. A better understanding of brain mechanisms and contributory stress would have an enormous impact on the public's understanding of the vulnerabilities for these disorders, influence medical and legal response to these problems, could lead to a new understanding of these phenomena, and stimulate a better means of prevention and treatment.

ELIGIBILITY:
Inclusion Criteria:

1. age 18-50 years inclusive;
2. able to read and write English;
3. for women, being in follicular phase of menstrual cycle at the time of the PET scan as determined by calculating the time since the last menses and assessments of serum hormone levels;
4. 30 < BMI < 35 for obese subjects (upper limit of 35 selected given our experience with heavier individuals fitting comfortably in the MRI scanner) and 18.5 < BMI <25 for normal weight subjects, and no recent weight changes in prior 12 weeks prior to the study;
5. for alcohol dependent patients meet current DSM-IV criteria for alcohol dependence or being in partial remission; abstinence on the MRI and PET scan days will be determined by patient self-report, breath alcohol tests (BACs) conducted during inpatient stay at the CNRU/GCRC, participants have to be non-obese BMI < 30, and
6. for current daily smokers, having smoked 10 or more cigarettes daily for the past year and CO level > 10 ppm at intake; for non-smokers, no tobacco consumption for more than one year and never having used tobacco daily.

Exclusion Criteria:

1. any major neurological illness or injury and any current or prior clinically significant mental health or substance use disorder (with possible exception of nicotine dependence and alcohol dependence per the inclusion criteria) as determined by SCID interview and the judgement of the PI;
2. use of any psychoactive medication within past three weeks;
3. any significant unstable medical condition such as asthma or heart disease which may limit the interpretation of the imaging results, for example due to changes in tracer delivery in hypertensive patients;
4. IQ<70 based on past intelligence testing;
5. any metal in body that would pose a risk with MRI; and
6. claustrophobia that would interfere with MRI or PET imaging;
7. presence of alcohol and drug use in the 72 hours prior to scanning, with the exception of tobacco;
8. pregnancy or nursing for women,
9. peri- and post- menopausal women, and those with ovarectomies will be excluded
10. current eating disorders, including binge eating.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 24 unmedicated abstinent alcohol dependent patients, 24 obese individuals and 24 individually matched healthy control subjects
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2007-07; Primary Completion 2012-07 (Actual); Study Completion 2023-01-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc N Potenza, MD, PhD, Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States